CLINICAL TRIAL: NCT04053803
Title: An Open-label Extension Study of IMR-687 in Adult Patients With Sickle Cell Anemia (Homozygous HbSS or Sickle-β0 Thalassemia) Who Participated in Study IMR-SCD-102
Brief Title: An Extension Study of IMR-687 in Adult Patients With Sickle Cell Anemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imara, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMR-SCD-102-EXT; 2018-003805-25 (EudraCT Number)
Record Dates: First submitted 2019-07-18; First posted 2019-08-13 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: IMR-687

INTERVENTIONS:
Drug: IMR-687 — Oral administration of once daily IMR-687

SUMMARY:
This is an open-label extension study of IMR-687 in adult patients who completed Imara's blinded Phase 2a study (IMR-SCD-102). The open-label extension study will evaluate long-term safety and tolerability.

DETAILED DESCRIPTION:
This is an open-label extension study of IMR-687 in adult patients with SCA who were previously participants in the Phase 2a study titled "A Phase 2a, Randomised, Double-Blind, Placebo-Controlled Study of IMR-687 in Adult Patients with Sickle Cell Anaemia (Homozygous HbSS or Sickle-β0 Thalassemia)."

This open-label extension study with IMR-687 will evaluate the long-term safety and tolerability of IMR 687 in adult SCA patients. Exploratory long-term PD parameters will also be examined.

ELIGIBILITY:
Inclusion Criteria:

1. Completed Study IMR-SCD-102.
2. Female subjects must not be pregnant, not be breast feeding, and be highly unlikely to become pregnant. Male subjects must be unlikely to impregnate a partner.
3. Subjects must be capable of giving informed consent and reading and signing the informed consent form after the nature of the study has been fully explained to them
4. Subjects must be willing and able to complete all study assessments and procedures and to communicate effectively with the investigator and site staff.

Exclusion Criteria:

1. Subjects with Hb >12.5 g/dL or <6 g/dL
2. Subjects with known active hepatitis B or hepatitis C, with active or acute event of malaria or who are known to be positive for human immunodeficiency virus (HIV)
3. eGFR <50 mL/min
4. AST/ALT > 3x the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with adverse events and serious adverse events | Baseline to Month 49
  1. Incidence of Adverse Events
  2. Incidence of Serious Adverse Events
Proportion of patients with changes in safety cardiac parameters | Baseline to Month 49
  a. Changes in 12-lead ECG parameters that are clinically significant and measured in milliseconds (ms).
  The parameters are: PR interval, QRS duration, QT interval, ST segment duration and T wave duration.
Proportion of patients with changes in clinical laboratory tests | Baseline to Month 49
  a. Clinically significant changes in clinical laboratory tests including serum chemistry, serum hematology and urinalysis
Proportion of patients with clinically significant abnormal vital signs | Baseline to Month 49
  1. Blood pressure measured in mmHg
  2. Pulse measured in beats per minute
  3. Respiration rate measured in breaths per minutes
  4. Temperature as measured in degrees F0 or C0

CONTACTS AND LOCATIONS:
Overall Officials: Karen Tang, MD, Study Director — Imara, Inc.
Locations (7):
- United States (3):
  - University of Connecticut Health Center, Farmington, Connecticut
  - Foundation for Sickle Cell Disease Research, Hollywood, Florida
  - Baylor Scott & White Medical Center - Temple, Temple, Texas
- United Kingdom (4):
  - Bristol Haematology and Oncology Centre, Bristol
  - University College London Hospital NHS Foundation Trust, London
  - Guy's and St Thomas Hospital CRF, London
  - Royal London Hospital, London